CLINICAL TRIAL: NCT02555774
Title: A Prospective, Three-arm, Parallel Design, Controlled Trial to Assess Efficacy of Cognitive Training in Subjective Memory Impairment
Brief Title: Efficacy of Cognitive Training in Subjective Memory Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jae-Hong Lee, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YJeongHong
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Memory Loss
Keywords: subjective memory impairment; cognitive training
MeSH Terms: conditions — Memory Disorders | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- cognitive training (Experimental): Cognitive training programs 2 times a week for 3 months (totally 24 sessions) for 90 minutes per session. Lifestyle modification is educated first, then weekly phone call for lifestyle modification is done by investigators.
  Interventions: Behavioral: cognitive training; Behavioral: lifestyle modification
- lifestyle modification (Active Comparator): This group receives only lifestyle modification for 3 months. Lifestyle modification is educated at the first, then weekly phone call for lifestyle modification is done by investigators. The method of lifestyle modification is same with the first arm.
  Interventions: Behavioral: lifestyle modification
- No intervention (No Intervention): This group receives no intervention.

INTERVENTIONS:
Behavioral: cognitive training — cognitive training is held 2 times a week for 3 months, 90 minutes per 1 session. It includes cognitive exercise of multiple cognitive domains such as memory, attention, calculation, executive function and visuospatial function.
  Arms: cognitive training
Behavioral: lifestyle modification — education about lifestyle modification is done by investigators at the first day of the trial and the investigators conduct weekly phone call to participants to educate the lifestyle modifications
  Arms: cognitive training; lifestyle modification

SUMMARY:
This study evaluates the efficacy of cognitive training in subjects with subjective memory impairment. The first group will receive cognitive training and lifestyle modification in combination, the second group will receive only lifestyle modification, and the third group will receive no intervention.

DETAILED DESCRIPTION:
Subjective memory impairment is currently thought to be a risky state of progression to Alzheimer's disease. This study aims to confirm whether cognitive training in subjective memory impairment would show improvement in the subjective and objective cognition. We include subjects with normal cognition but complained subjective feeling of memory decline and conduct cognitive training programs combined with lifestyle modifications for 3 months. We evaluate the neuropsychological tests and questionnaires about subjective improvement after 3 months of interventions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who showed normal range (above 16percentile of norm) in all domains of detailed neuropsychological tests battery named Seoul Neuropsychological Screening Battery (SNSB)
* Clinical dementia rating (CDR) score of 0
* Subjects with at least 3 years of formal education

Exclusion Criteria:

* Subjects with mild cognitive impairment or dementia
* Subjects who was diagnosed as any neurological disorders such as epilepsy, stroke, hemorrhage, hydrocephalus, Parkinson's disease or brain tumor
* Subjects with uncontrolled severe medical conditions according to investigator's opinion

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Paired associates learning test | 3 month
  paired associates learning test is a part of computerized neuropsychological tests battery named CANTAB (Cambridge Neuropsychological Test Automated Battery). The scores are shown as total number of errors.
Rapid visual information processing test | 3 month
  rapid visual information processing is a part of computerized neuropsychological test battery named CANTAB. The score is shown as correct response rate.%
Pattern recognition memory test | 3 month
  paired associates learning test is a part of computerized neuropsychological tests battery named CANTAB (Cambridge Neuropsychological Test Automated Battery). The score is shown as correct response rate.%
Spatial working memory test | 3 month
  paired associates learning test is a part of computerized neuropsychological tests battery named CANTAB (Cambridge Neuropsychological Test Automated Battery). The scores are shown as total number of errors.

SECONDARY OUTCOMES:
cognitive failure questionnaire | 3 month
  questionnaire for measuring self reported cognitive status. score range: 0-100. Higher score means worse cognitive status.
Mini-mental state examination | 3 month
  mini-mental state examination that examines general cognition. range 0-20. Higher score means better cognition.
Geriatric depression scale | 3 month
  questionnaire for depression measuring. score range:0-15. lower score means less depression.
Beck anxiety index | 3 month
  questionnaire for self reporting anxiety measuring. range:0-63. low score means less anxiety.
Seoul instrumental activities of daily living | 3 month
  scale for measuring activities of daily living limitation. score range 0-45. low score means better ability.
Rey complex figure copy test | 3 month
  test for visuospatial function. Participants should copy the complex figure. score range: 0-36. Higher score means better visuospatial function.
Digit symbol test | 3 month
  a test for attention and psychomotor speed. Participants are instructed to write an appropriately matched code for each number. Correct number is counted. score range: 0-76. Higher score means better function.
Seoul verbal learning test, immediate recall | 3 month
  measuring tool for immediate memory function. Investigators read 12 words to participants. Participants should remember the words. Tests are done 3 times. score range: 0-36. Higher score means better immediate memory function
Seoul verbal learning test, delayed recall | 3 month
  measuring tool for 20 minutes delayed memory function. After 20 minutes from the immediate recall test, participants should remember the words. score range: 0-12. Higher score means better delayed memory function
Seoul verbal learning test, delayed recall | 3 month
  measuring tool for cued recall of verbal memory function. score range: 0-24. 2. Higher score means better memory recognition function
Logical memory test, delayed recall | 3 month
  logical memory test is a part of a neuropsychological test named Wechsler

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Hong Lee, MD,PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Jae-Hong Lee, Seoul, South Korea